CLINICAL TRIAL: NCT07333001
Title: Efficacy and Safety of 7-day Triple Therapy Containing Amoxicillin and Tetracycline Versus 14-day Dual Therapy for Helicobacter Pylori Eradication
Acronym: PSM
Status: Completed | Type: Observational
Sponsor: Yueyue Li (Other)
Collaborators: Qilu Hospital of Shandong University (Other)
Responsible Party: Sponsor-Investigator, Yueyue Li, Associate Professor, Qilu Hospital of Shandong University
Organization: Qilu Hospital of Shandong University (Other)
Other Study IDs: 202512
Record Dates: First submitted 2025-12-27; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: HELICOBACTER PYLORI INFECTIONS
Keywords: Helicobacter pylori; triple therapy; dual therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- triple therapy
  Interventions: Drug: 7-day triple therapy
- dual therapy
  Interventions: Drug: 14-day dual therapy

INTERVENTIONS:
Drug: 7-day triple therapy — vonoprazan 20 mg twice daily, amoxicillin 1000 mg twice daily, and tetracycline 500 mg four times daily for 7 days
  Groups: triple therapy
Drug: 14-day dual therapy — vonoprazan 20 mg twice daily and amoxicillin 1000 mg three times daily for 14 days
  Groups: dual therapy

SUMMARY:
With the increasing prevalence of antibiotic resistance, the clinical efficacy of conventional 7-day triple therapy for Helicobacter pylori eradication has been substantially diminished. However, the efficacy and safety of a 7-day triple regimen based on amoxicillin and tetracycline warrant further investigation. This retrospective study was designed to compare the efficacy and safety of a 7-day triple therapy based on amoxicillin and tetracycline combination versus the standard 14-day high-dose dual therapy for H. pylori infection. Data on therapies for H. pylori eradication were extracted between January 2023 and October 2025 at Qilu Hospital of Shandong University. Two regimens were compared based on 1:3 propensity score matching: 7-day triple therapy (vonoprazan 20 mg twice daily, amoxicillin 1000 mg twice daily, and tetracycline 500 mg four times daily) and 14-day high-dose dual therapy (vonoprazan 20 mg twice daily and amoxicillin 1000 mg three times daily). Eradication rates and incidence of adverse events were assessed.

ELIGIBILITY:
Inclusion Criteria:

* patients aged 18-70 years;
* patients with H. pylori infection confirmed by 13C/14C-urea breath test or rapid urease test;
* patients with no history of H. pylori eradication therapy

Exclusion Criteria:

* patients with severe underlying diseases, such as hepatic insufficiency, renal insufficiency, immunosuppression, malignant tumors, and coronary heart disease;
* patients with active gastrointestinal bleeding;
* patients with a history of upper gastrointestinal surgery;
* patients allergic to treatment drugs;
* patients with medication history of bismuth, antibiotics within 4 weeks, or proton pump inhibitors within 2 weeks;
* patients who were pregnant or lactating or unwilling to take contraceptive measures during the trial;
* patients with other behaviors that may increase the risk of disease, such as alcohol and drug abuse;
* incomplete data.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * patients aged 18-70 years;
  * patients with H. pylori infection confirmed by 13C/14C-urea breath test or rapid urease test;
  * patients with no history of H. pylori eradication therapy
Sampling Method: Non-Probability Sample
Enrollment: 508 (Actual)
Dates: Start 2025-11-01 (Actual); Primary Completion 2025-12-15 (Actual); Study Completion 2025-12-27 (Actual)

PRIMARY OUTCOMES:
eradication rate | six weeks after treatment

SECONDARY OUTCOMES:
incidence of adverse events | immediately after treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Qilu Hospital of Shandong University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No